CLINICAL TRIAL: NCT06151951
Title: Comparative Effects of Visual and Pressure Biofeedback on Pain, Range of Motion and Disability in Symptomatic Forward Head Posture.
Brief Title: Comparative Effects of Visual and Pressure Biofeedback in Symptomatic Forward Head Posture.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0154
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Forward Head Posture
Keywords: FHP

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Movement control training of Neck flexor muscles with Pressure Biofeedback along with baseline treatment
  Interventions: Other: Cervical Stabilization; Device: Pressure Biofeedback
- Group B (Experimental): Movement control training of Neck flexor muscles with Visual Biofeedback along with baseline treatment
  Interventions: Other: Cervical Stabilization; Device: Visual Biofeedback

INTERVENTIONS:
Other: Cervical Stabilization — Isometric stretching and strengthening exercises of Neck flexor muscle including suboccipitalis, levator scapulae,scalnae anterior and upper trapezius. Each exercise hold for 6 second and then release and repeated 10 times respectively 3 times in a week for 4 weeks. Therefore, the total exercise time will be 5-10 mints.
Device: Pressure Biofeedback — In this method patients in supine position. Sphygmomanometer is used and 100 mmHg pressure will be maintained before the treatment start then cuff will be placed under the occiopit of spine and patient will be asked to press the cuff against the occiopit until gauze show target pressure then hold this position for 6 second and release. Repeated this pressure to 10 times, 3 times in a week for 4 weeks. Therefore, the total exercise time will be 5-10 mints.
  Baseline Treatment
  Before starting the session participants received moist heat pack and soft tissue massage on cervical for 10 to 15 mints followed by movement control training.
  Arms: Group A
Device: Visual Biofeedback — In this method Led Head Band light will be used as a visual feedback. Patients in sitting or standing position with neck straight with the alignment of front wall marking followed by control movement training. Patient will be asked to follow the marking through head band light while performing motion control training. Each exercise hold for 6 second and then release and repeated 10 times respectively 3 times in a week for 4 weeks. Therefore, the total exercise time will be 5-10 mints.
  Baseline Treatment
  Before starting the session participants received moist heat pack and soft tissue massage on cervical for 10 to 15 mints followed by movement control training.
  Arms: Group B

SUMMARY:
This study aims to determined the comparative effect of visual and pressure biofeedback on Pain,Disability and Range of Motion in young and middle aged adults diagnosed with forward head posture.

DETAILED DESCRIPTION:
Forward head posture describes the shifting of the head forward with the chin poking out. It is caused by increased flexion of the lower cervical spine and upper thoracic.

Forward head posture is the most frequently observed postural deviations and is said to be associated with shortening of posterior cervical extensors and weakening of the anterior deep cervical flexors. In this randomized control trial participants showing forward head posture will be randomly assigned into two intervention groups. 28 subjects were divided equally into two groups 14 each containing both genders. Group A (Experimental group) will be given isometric strengthening and stretching training guided pressure biofeedback.

Group B (Experimental group) will be given isometric strengthening and stretching training of deep cervical flexor (DCF) muscle guided through visual biofeedback .

Each participant will be receive a total of twelve treatment sessions over a four-week period. The efficacy of the interventions will be assessed at the beginning (first session) and conclusion (last session) of the treatment period. The assessment will encompass various outcome measures. Pain intensity will be evaluated using the Numeric Pain Rating Scale (NPRS), while disability levels will be measured using the Neck Disability Index (NDI). The cervical active range of motions (CAROMs) will be assessed by goniometry. Finally, the visual feedback referred as indicator of measuring forward head posture by evaluating these outcome measures insights will be gained into the impact of the interventions on the participants' symptoms and postural alignment through light. The randomized design of the trial provide valuable information to healthcare professionals on how to manage symptomatic forward head posture and may contribute to the development of future research in this area.

ELIGIBILITY:
Inclusion Criteria:

1. Participants would be complaining of neck pain as a primary complain and age of 20- 35 year was recruited in the study .

2 . Male and female both gender are included in the study.

3. patient with Craniovertebral angle (CVA)<53 degree were included in the study .

4. Score more than 3 on NPRS and more than 10 on NDI.

Exclusion Criteria:

Participant failing to fall in this category would be excluded of the study.

1. Neurogenic findings like cervical trauma, myopathy, vestibular pathology, dizziness, visual problem, spinal Fracture, dislocation and hypertension will not include in the study.
2. History of sever metabolic diseases.
3. History of recurrent surgery in upper thoracic and lumber vertebrae
4. History of recent fractures in shoulder and neck region.
5. History of tumor. -

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks
  The NPRS is a subjective pain rating scale using an 11-point scale from 0 to 10, where 0 means 'no pain' and 10 means 'intolerable pain'. Participants select the whole number that best represents their level of pain. The reliability is >0.95 with ICC values 0.86- 0.95
Neck Disability Index (NDI) | 4 weeks
  NDI is a self-reported questionnaire which is formulated to assess pain that restricts the activities of daily living (ADL); it also helps to determine self-assessed disability. NDI has 10 domains covering pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Scores range from 0 to 50, with 50 being the greatest levels of dysfunction. It is a valid and reliable tool with ICC=0.98
Pressure Biofeedback (Simple Sphygmomanometer) | 4 weeks
  It is used to measure the neck muscle strength. It was consisting of 3 chamber air filled pressure bag, a catheter & sphygmomanometer gauze. To measure the strength, cuff is placed under occipital in supine position for Neck flexor and under forehead in prone position for neck extensor muscle. After setting pressure with the baseline Pressure of 100 mmHg, patient was asked to put maximum effort on cuff by giving 6 seconds hold for 3 repetitions. After taking the mean value, it is compared with the normal extensor flexor.

SECONDARY OUTCOMES:
Visual Biofeedback (LED Headband light) | 4 weeks
  This light is known as light panel that contain rectangular shape light focusing panel that maintain the focus through manual adjustment.
goniometry | 4 weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position. In orthopedics, the former description applies more. It is valid and reliable tool for measuring range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, Principal Investigator — Riphah International University; Nusrat Prveen, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Bahawal Victoria Hospital QAMC Bahawalpur, Bahawalpur, Punjab Province
  - Bahawal Victoria Hospital QAMC Bahawalpur, Chak Four Hundred Fifty-four, Punjab Province

IPD SHARING:
Plan to Share IPD: No